CLINICAL TRIAL: NCT06208826
Title: A Single-center Phase II Study to Investigate the Immune Maintenance Therapy Pattern in Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma Who Have Achieved MPR After Neoadjuvant Immunotherapy Combined With Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FERRY
Record Dates: First submitted 2024-01-07; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — toripalimab; Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toripalimab (Experimental): toripalimab, IV, 240mg, q3w, for 15 cycles
  Interventions: Drug: Toripalimab
- SOC CCRT or radiotherapy (Active Comparator): Standard concurrent radiochemotherapy or postoperative radiotherapy
  Interventions: Radiation: Radiation Therapy; Drug: Cisplatin

INTERVENTIONS:
Drug: Toripalimab — Toripamab, IV, 240mg, every 3 weeks for 15 cycles
  Arms: Toripalimab
Radiation: Radiation Therapy — Radiation Therapy
  Arms: SOC CCRT or radiotherapy
Drug: Cisplatin — Chemotherapy agent
  Arms: SOC CCRT or radiotherapy

SUMMARY:
Head and neck cancer is the malignant tumor with the highest morbidity and mortality, of which 60% present with locally advanced disease at initial diagnosis, and the 5-year survival rate of standard treatment is less than 30%. Standard of care (SOC) including adjuvant and neoadjuvant therapy can provides only about 5-10% clinical benefit. According to the available data on the application of immunotherapy as adjuvant therapy in operable patients, adjuvant immunotherapy is safe and feasible, with a significant trend of benefit. Based on the above positive and meaningful clinical needs and scientific basis, it is very necessary to carry out clinical trials of adjuvant immunotherapy. The primary objective of this study is to evaluate the efficacy and safety of immune maintenance therapy in patients with locally advanced head and neck squamous cell carcinoma who achieve MPR after neoadjuvant immunotherapy combined with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to give an informed consent for the study.
* Males or females aged 18 to 80 years.
* Have an Eastern Co-operative Oncology Group (ECOG) performance status less than equal to 1.
* Pathologically (histologically or cytologically) confirmed, non-metastatic diagnosis of squamous cell carcinoma of head and neck (SCCHN).
* Achievement of major pathological reaponse (MPR) after surgery with neoadjuvant immunotherapy combined chemotherapy.
* Adequate bone marrow, liver, and renal function:

Absolute neutrophil count ≥ 1.5 × 10^9/L, hemoglobin ≥ 9.0g/dL, platelets ≥100000/μL; ALT and AST < 2.5× upper limit of normal (ULN), total bilirubin ≤ 1.5×ULN； Creatinine clearance ≥ 60 ml/min； APTT≤ 1.5×ULN.

Exclusion Criteria:

* Participant has metastatic/unresectable SCCHN.
* Have an active autoimmune disease requiring systemic treatment or a documented history of clinically severe autoimmune disease.
* With active hepatitis B or C, or known history of positive HIV test, or acquired immunodeficiency syndrome.
* With interstitial pneumonitis, non-infectious pneumonitis, active pulmonary tuberculosis, or history of pulmonary tuberculosis infection that were not controlled by treatment.
* With active infection requiring systemic therapy.
* Received any investigational drug within 4 weeks prior to the first dose, or concurrently enrolled in another clinical trial.
* Any other factors that are not suitable for inclusion in this study judged by investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | up to 4 years
  defined as the time from random assignment to documented local or regional relapse, distant metastasis, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Over survival (OS) | up to 4 years
  OS is defined as the time from randomization to death due to any cause or censored at the date of last follow-up.
Toxicity Adverse events | up to 1 year
  Grade 1-5 AEs according to NCI-CTCAE V5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No